CLINICAL TRIAL: NCT04290260
Title: Randomized Controlled Trial of the Effectiveness of Bra Application in Women as a Device for Prevention of Surgical Wound Dehiscence in the Post-operative Cardiac Surgery
Brief Title: Use of the Bra as Prevention of Sternal Wound Dehiscence in Cardiac Surgery
Acronym: DEHISCENCIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundació Institut Germans Trias i Pujol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AC-14-060; PR-1850/14 (Other Grant/Funding Number: Col·legi Oficial d'Infermeres i Infermers de Barcelona)
Record Dates: First submitted 2019-12-03; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Cardiac Surgical Procedures; Wound Healing
Keywords: Cardiovascular nursing; Bra; Dehiscence; Sternotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of breast bra (Experimental): Patients allocated on this group wear a breast bra from admission to hospital discharge.
  Interventions: Other: Use of breast bra
- Usual care (Active Comparator): Usual care: participants will not wear a breast bra until discharge from the hospital
  Interventions: Other: Usual care (not use of bra)

INTERVENTIONS:
Other: Use of breast bra — Patients will use a breast from admission to hospital discharge
  Arms: Use of breast bra
Other: Usual care (not use of bra)
  Arms: Usual care

SUMMARY:
The aim of the study was to assess the efficacy of bra application as a prevention of dehiscence in women with median sternotomy.

DETAILED DESCRIPTION:
Background: it is known that the size and support of the breasts are a specific problem in post-operative women of cardiac surgery by means of medium sternotomy. There is little evidence of the therapeutic action of the bra as a measure to prevent dehiscence of the surgical wound.

Aim: To assess the efficacy of bra application as a prevention of dehiscence in women with median sternotomy.

Methods: Randomised clinical trial; post-test control group in women undergoing cardiac surgery by mean sternotomy. Groups: application of post-surgical or non-surgical breast bra. Endpoint: incidence of dehiscence. Other variables: sociodemographic, signs of infection, pain, related to assessment of the wound on admission. Assessment of the surgical wound daily, at discharge, at month, 3 months and 6 months post discharge.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Cardiac surgery intervention in the Germans Trias i Pujol University Hospital with non-critical preoperative
* Surgical intervention performed throughout medium sternotomy

Exclusion Criteria:

* More than 72 hours admitted in an intensive care unit after surgery
* Cognitive impairment or severe physical disability
* Mastectomy
* External wound occlusion with Opsite® fixative absorbent dressing
* Emergency surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Dehiscence | Baseline (admission) to 6 months after hospital discharge
  Dehiscence in the surgical wound. Criteria defined according to an established scale for the assessment of surgical wounds contemplated in the GacelaCare® computer system used in Germans Trias i Pujol University Hospital. Values may be "Yes" or "No".

CONTACTS AND LOCATIONS:
Overall Officials: Violeta Díaz Herrera, RN, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No